CLINICAL TRIAL: NCT05014100
Title: A Multicenter Clinical Study of Orelabrutinib Combined With Lenalidomide and Rituximab (OR2) in the Treatment of Recurrent and Refractory CD20+ B-cell Lymphoma
Brief Title: Orelabrutinib in Combination With R2 Regimen for R/R CD20+ B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Puyang Oilfield General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PYOFGHhema001
Record Dates: First submitted 2021-07-29; First posted 2021-08-20 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — orelabrutinib; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The treatment group (Experimental): Orelabrutinib 150mg once daily in a 28-day cycle. Lenalidomide 25mg once daily for 21 days and rituximab 375mg/m2 for 7 days
  Interventions: Drug: Orelabrutinib tablet; Drug: Lenalidomide

INTERVENTIONS:
Drug: Orelabrutinib tablet — Subjects received orelabrutinib150mg orally once daily for a 28-day cycle. Throughout the study period, all subjects continued treatment until one of the following conditions occurred: disease progression, intolerable toxicity, death, withdrawal of informed consent, or loss of follow-up
Drug: Lenalidomide — Lenalidomide 25mg once daily for 21 days and rituximab 375mg/m2 for 7 days
  Throughout the study period, all subjects continued treatment until one of the following conditions occurred: disease progression, intolerable toxicity, death, withdrawal of informed consent, or loss of follow-up
  Other Names: RR

SUMMARY:
Obrutinib is a highly selective BTKi and has shown efficacy in CLL/MCL. This study aims to investigate the initial efficacy and safety of obrutinib combined with R2 regimen in the treatment of relapsed or refractory CD20+B cell lymphoma

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (BTK), a member of the TEC family of non-receptor tyrosine proteins, is expressed in B lymphocytes, mast cells, macrophages, monocytes, neutrophils, etc., and is a key molecule in the signaling of B cell antigen receptor (BCR). The development and differentiation of B cells can be controlled by activating positive cell cycle regulators and differentiated cytokines, and the survival and proliferation of B cells can be controlled by regulating the expression of pro-apoptotic and anti-apoptotic proteins. BTK inhibitors inhibit B cell maturation and activation by targeting the BCR signaling pathway.

Compared with other BTK inhibitors, orelabrutinib is highly selective. Previous studies showed that among 456 tested kinases, the inhibition rate of orelabrutinib only exceeded 90% at 1µM concentration, which is the BTK inhibitor with the highest kinase selectivity reported so far. It has shown a good safe treatment window in animal models, and its pharmacokinetic properties are far superior to those of ibrutinib.

In the Phase I dose exploration study of orelabrutinib in Australia, the single dose was from 20mg/ day to 400mg/ day, and the continuous dose was from 100mg/ day to 200mg/ day. No serious adverse events related to the drug occurred, and no dosion-limiting toxicity was found. The main adverse reactions were headache, intubation pain, fatigue, etc. Most of them were mild and generally well tolerated, providing a reference for the selection of subsequent clinical drug dosage.

Phase I/II clinical trials of orelabrutinib for MCL and CLL/SLL have been conducted in more than 20 centers across the country. Based on preliminary results observed in Phase I, obrutinib has demonstrated excellent safety and tolerability in patients with relapsed refractory MCL and CLL/SLL. Most of the adverse reactions were grade 1-2. Good results have been observed early on in patients. Good pharmacokinetic/pharmacokinetic properties.

Several studies have shown that ibrutinib combined with lenalidomide and rituximab improves survival in patients with relapsed refractory diffuse large B-cell lymphoma. In addition, ibrutinib combined with lenalidomide and rituximab has been included in the expert recommendation of multiple relapsed and refractory B-cell lymphomas in the 2021CSCO Lymphoma Guidelines.

In conclusion, orelabrutinib and lenalidomide combined with rituximab demonstrated good efficacy and tolerability in the treatment of relapsed refractory B-cell lymphoma. Moreover,orelabrutinib has better selectivity than ibrutinib, so we believe that orelabrutinib combined with lenalidomide and rituximab (OR2) may have better efficacy in the treatment of relapsed and refractory B-cell lymphoma, and there is no research report on this regimen. The application of this regimen may bring new hope for relapsed refractory B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years old, ≤75 years old, gender is not limited;

  2) CD20+B cell lymphoma was confirmed by histopathology, with at least one intranode lesion larger than 1.5CM in length and extranodal lesion larger than 1.0CM in diameter.

  3) Patients with recurrent or refractory CD20+ B-cell lymphoma who have previously received ≥1 line and ≤5 line of different chemotherapy and/or targeted drug therapy failure and lack effective and standard treatment options;

  4) ECOG strength score 0-2;

  5) Medical records that have failed to respond to the latest systematic treatment (not reaching CR/PR) or disease progression after remission;

  6) Major organ functions meet the following criteria:

A) Blood routine: neutrophils absolute value ≥1.5×109/L, platelets ≥75×109/L, hemoglobin ≥75g/L; Absolute neutrophils if associated with bone marrow invasion

≥1.0×109/L, platelet ≥50×109/L, hemoglobin ≥75g/L;

B) Blood biochemistry: total bilirubin ≤1.5 times ULN, AST or ALT≤3 times ULN; Serum creatinine ≤1.5 ULN; Serum amylase ≤ULN;

C) Coagulation function: International standardized ratio (INR) ≤1.5 times ULN.

7) Expected survival ≥3 months;

8) Voluntarily sign written informed consent before screening.

Exclusion Criteria:

* 1) Current or previous malignancy, unless radical therapy has been performed and there is no evidence of recurrence or metastasis in the past 5 years;

  2) Non-hematologic toxicity of previous antitumor therapy did not return to ≤ grade 1 (excluding hair loss)

  3) Have uncontrolled or significant cardiovascular disease

  7) Had active bleeding within 2 months prior to screening, or was taking anticoagulant drugs, or was considered by the investigator to have a clear tendency to bleeding;

  (8) Urine protein ≥2+, and 24 h urine protein quantification ≥ 2G /24 h;

  9) History of deep vein thrombosis or pulmonary embolism;

  10) The toxicity of the pre-screening treatment regimen has not recovered, and there are still toxicity reactions above grade 1;

  11) Subjects with clinically significant gastrointestinal abnormalities that may affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy;

  12) A history of organ transplantation or allogeneic bone marrow transplantation;

  13) Major surgery or minor surgery within 6 weeks prior to screening or 2 weeks prior to screening. Major surgery is surgery performed under general anesthesia, but endoscopic examination for diagnostic purposes is not considered major surgery. Insertion of vascular access devices will be exempt from this exclusion criterion;

  14) Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C virus infection (positive results by POLYMERase chain reaction [PCR]).

  15) Current subjects with pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of lung function;

  16) Suitable and ready for stem cell transplantation;

  17) Any mental or cognitive impairment that may limit his/her understanding, implementation and compliance with the informed consent;

  18) Subjects with drug and alcohol abuse;

  19) Pregnant and lactating women and subjects of childbearing age who do not want to take contraceptive measures;

  20) Combined with drugs with moderate to severe inhibitory effect or strong induction effect on cytochrome P450 CYP3A;

  21) Other conditions that the researcher considers unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Enrollment to the last patient complete 6cycles（each cycle is 28 days）, an average of 1 year
  The proportion of patients receiving a OR2 regimens who are in remission

CONTACTS AND LOCATIONS:
Overall Officials: Xuejun Guo, PHD, Principal Investigator — Puyang Oilfield General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ujjani C, Wang H, Skarbnik A, Trivedi N, Ramzi P, Khan N, Cheson BD. A phase 1 study of lenalidomide and ibrutinib in combination with rituximab in relapsed and refractory CLL. Blood Adv. 2018 Apr 10;2(7):762-768. doi: 10.1182/bloodadvances.2017015263. PMID 29610115
- [Background] Ujjani CS, Jung SH, Pitcher B, Martin P, Park SI, Blum KA, Smith SM, Czuczman M, Davids MS, Levine E, Lewis LD, Smith SE, Bartlett NL, Leonard JP, Cheson BD. Phase 1 trial of rituximab, lenalidomide, and ibrutinib in previously untreated follicular lymphoma: Alliance A051103. Blood. 2016 Nov 24;128(21):2510-2516. doi: 10.1182/blood-2016-06-718106. Epub 2016 Oct 3. PMID 27697771
- [Background] Goy A, Ramchandren R, Ghosh N, Munoz J, Morgan DS, Dang NH, Knapp M, Delioukina M, Kingsley E, Ping J, Beaupre DM, Neuenburg JK, Ruan J. Ibrutinib plus lenalidomide and rituximab has promising activity in relapsed/refractory non-germinal center B-cell-like DLBCL. Blood. 2019 Sep 26;134(13):1024-1036. doi: 10.1182/blood.2018891598. Epub 2019 Jul 22. PMID 31331917
- [Background] Yu H, Wang X, Li J, Ye Y, Wang D, Fang W, Mi L, Ding N, Wang X, Song Y, Zhu J. Addition of BTK inhibitor orelabrutinib to rituximab improved anti-tumor effects in B cell lymphoma. Mol Ther Oncolytics. 2021 Apr 3;21:158-170. doi: 10.1016/j.omto.2021.03.015. eCollection 2021 Jun 25. PMID 33981831